CLINICAL TRIAL: NCT03437057
Title: Maintenance of an Antiaggregation by Acetylsalicylic Acid, Less or Equal to 250mg While a Extracorporeal Lithotripsy (ECL) Session on a Kidney Stone is Perfomed: Comparative Unicentric Prospective Study
Brief Title: Maintenance of an Antiaggregation by Acetylsalicylic Acid, While a Extracorporeal Lithotripsy Session on a Kidney Stone is Perfomed: Comparative Unicentric Prospective Study
Acronym: KARLITHO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RBHP_2017_GUANDALINO; 2017- A01453-50 (Other: ANSM)
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Renal Lithiasis; Antiplatelet; Hematoma
Keywords: ECL; Hematoma; Antiplatelet
MeSH Terms: conditions — Nephrolithiasis; Hematoma | interventions — Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with acethylsalicylic acid 250 mg (Experimental): Prospective single-arm study to estimate the risk of renal hematoma when performing a session of lithotripsy for renal lithiasis, on a 15-day scanner, in patients treated with acetylsalicylic acid not suspended.
  Interventions: Other: acetylsalicylic acid (below or equal to) 250 mg

INTERVENTIONS:
Other: acetylsalicylic acid (below or equal to) 250 mg — Prospective single-arm study to estimate the risk of renal hematoma when performing a session of lithotripsy for renal lithiasis, on a 15-day scanner, in patients treated with acetylsalicylic acid not suspended.

SUMMARY:
Background/Rationale for the study:

Lithiasis pathology is increasingly common because of the change in our lifestyle and our food. Thus, we hold a prevalence for urinary lithiasis 10% in France currently including 13% of the male population and 6% of the female population.

The formation of urinary lithiasis is the result of a complex mechanism involving factors anatomical and infectious metabolics. They are classified according to their size, topography and composition.

The treatment of urinary lithiasis has changed dramatically in recent years. The recommendations of the French Urology Association (AFU) for the management of kidney stones and ureteral of the adult of 2004 give a certain place to the treatment by extracorporeal lithotripsy (ECL).

The ELC is indicated for the first purpose for lithiasis ureteral or renal lithiasis of less than 20 mm, whether or not associated with the setting up of a JJ stent. For kidney stones of more than 20 mm or complex or Coralliformes, the ECL can be associated with treatment with percutaneous nephrolithotomy. In addition, the ECL is indicated in case of residual cholelithiasis 3 months after a first treatment whatsoever.

It is found, as the main complication of the ECL, a risk of the appearance of Hematomas under capsular, peri-renal and intra-parenchymatous. Its prevalence is estimated to be between 6.2% and 13% according to studies.

ACETYLSALICYLIC ACID less or equal to 250 mg is the usual dosage of aspirin (for the adult), the Marketing Autorisation recognises in secondary prevention after a first myocardial or cerebral ischemic attack related to atherosclerosis. It entrains a reduction mortality and morbidity of cardiovascular causes.

Acetylsalicylic acid is currently being stopped 5 to 7 days before the ECL. The interest of maintaining the Acetylsalicylic acid is:

* A simplification of the management of patients under on acetylsalicylic acid below (or equal to) 250 mg (No modification of Treatment to be implemented)
* A cardiovascular risk decreased by maintaining their initial treatment without any modification.

Main objective:

Evaluation of the proportion of renal hematoma during the production of Lithotripsy for renal lithiasis, on a 15-day scan, in patients under on acetylsalicylic acid below (or equal to) 250 mg not stopped

Secondary objectives:

Evaluation of the efficacy of treatment with lithotripsy (Stone free, fragments Minimal residuals) Evaluation of the proportion of hematuria macroscopic post lithotripsy in Patients under on acethylsalicylic acid not stopped. Evaluate the rate of post-ECL complications requiring treatment, Analgesic, obstructive pyelonephritis.

Evaluate post-ECL pain due to hematoma or lithiasis migration Evaluation of the evolution of renal function post session of Lithotripsy on the patients under acethylsalicylic acid not stopped.

Type of Study: Interventional study, prospective, mono centric, single-arm

DETAILED DESCRIPTION:
Before the ECL:

Patients will be recruited during the urology consultation prior to the lithotripsy for kidney stones Kidneys (JJ stent in place or not) using an uninjected abdominal-pelvic or ultrasound scanner Renal coupled to a AUSP (urinary tree without preparation). ECL is an Unbody method that allows the calculation to be fragmented using shock waves Generated by a lithotripter. It will be given to them, after explanation of this method by the doctor during the consultation, a AFU information sheet on the ECL explaining its steps, possible complications, its follow-up.

After checking the inclusion and non-inclusion criteria, patients will be programmed to ECL without prior stop of acethylsalicylic acid.

At the ECL session:

Evaluation of blood pressure before the session and at the end. Medical history and treatment will be notified in the patient file Verification of blood balance (coagulation, renal function) and urinary (BU and ECBU) Evaluation of pain by analog visual scale (AVS) before and during the session. Notification of possible symptoms (adverse reactions = AR) in the medical file. Prescription of analgesics as well as blood balance and revaluation scanner at D15 Taking a post-ECL appointment with the reference urologist at D23 (+-2days)

After the ECL session: 3-week post-ECL Consultation:

Pain Assessment (AVS) Evaluation of the effectiveness of the ECL (stone clearance)

Reading of the scanner performed at D15 in search of a hematoma "(the scanner will also be replayed from systematically by the prescriber or a urologist of the service looking for a hematoma and the level of efficacy of the ECL + control of the blood balance in search of a inflammatory/infectious/anemia/renal function Chronology of the essay:

Duration of study estimated at: 5 years Start date of study (first patient included): 01/2018 End Date (end of follow-up of the last patient of the study): 01/2023 Total duration of participation in the study for the patient: 5 to 6 weeks The end-of-study date shall be transmitted to the competent authority and the MPC within 90 days.

If the study is to stop prematurely, the information will be transmitted within a period of 15 days The competent authority and the MPC. Main judgement criterion: Proportion of patients with renal hematoma when performing of lithotripsy for renal lithiasis, on a 15-day scanner.

Number of topics: 300 based on a 4-step sequential plan of Fleming type

Inclusion criteria:

Patients over 18 years of age benefiting from the social security scheme Patients with at least one renal lithiasis requiring treatment with extracorporeal lithotripsy (ECL)

Non-inclusion criteria:

Coagulation disorder known or discovered on the pre-therapeutic balance sheet Associated anticoagulant therapy. Presence of another contraindications to the ECL.

Conduct of the study:

Study is carried out in current practice at the CHU of Clermont Ferrand in the Department of Urology.

The patient will be seen in consultation by the urologist who shall prescribe the Lithotripsy sessions, inform him about the of the session and will provide him a AFU information sheet concerning the stages of the session, and then, prescribe a blood test to be presented to the lithotriptor on the day of the examination. Not additional accommodation to plan. The patient will return 3 weeks after the ECL session for his evaluation with the urologist. He will have previously completed a blood check and a 15-day scan of the lithotripsy session (instead of about 3 weeks usually).

Benefits and risks of this study:

Simplify patient management under acethylsalicylic acid. Decrease in cardiovascular risk by maintaining the acethylsalicylic acid. Increase of the risk of post-ECL hematoma

ELIGIBILITY:
Inclusion Criteria

* Over 18 yo patients
* Patients with 1 renal lithiasis (at least) requiring treatment with extracorporeal lithotripsy
* Patients taking Kardégic 75 (monotherapy

Exclusion Criteria:

* Patients with known (or previously known) bleeding disorders on the pre-treatment assessment
* Patients with anticoagulant therapy or other anti-aggregating therapy (eg Kardegic at 75mg, AVK, NACO, LMWH, HNF, P2Y12 inhibitor)
* Patients with another contrindication to the ECL.
* Patients with prescription of more than the outset 1 ECL session
* Tutelage, curatorship, justice safeguarding, deprived of liberties, unaffiliated SS, impaired comprehension abilities, pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the proportion of renal hematoma during the production of Lithotripsy for renal lithiasis | at 15 days
  Evaluation of the proportion of renal hematoma during the production of Lithotripsy for renal lithiasis, on a 15-day scan, in patients under acetylsalicylic acid (below or equal to 250mg) not stopped

CONTACTS AND LOCATIONS:
Overall Officials: Marlène GUANDALINO, MD, Study Director — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Donsimoni R, Hennequin C, Fellahi S, Troupel S, Moel GL, Paris M, Lacour B, Daudon M. New aspects of urolithiasis in France. GERBAP: Groupe d'Evaluation et de Recherche des Biologistes de l'Assistance Publique des Hopitaux de Paris. Eur Urol. 1997;31(1):17-23. PMID 9032529
- [Background] Bihl G, Meyers A. Recurrent renal stone disease-advances in pathogenesis and clinical management. Lancet. 2001 Aug 25;358(9282):651-6. doi: 10.1016/S0140-6736(01)05782-8. PMID 11530173
- [Background] Daudon M, Dore JC, Jungers P, Lacour B. Changes in stone composition according to age and gender of patients: a multivariate epidemiological approach. Urol Res. 2004 Jun;32(3):241-7. doi: 10.1007/s00240-004-0421-y. Epub 2004 May 4. PMID 15127165
- [Background] Streem SB, Yost A, Mascha E. Clinical implications of clinically insignificant store fragments after extracorporeal shock wave lithotripsy. J Urol. 1996 Apr;155(4):1186-90. PMID 8632527
- [Background] Tolley DA. Consensus of lithotriptor terminology. World J Urol. 1993;11(1):37-42. doi: 10.1007/BF00182170. PMID 8490666
- [Background] Candau C, Saussine C, Lang H, Roy C, Faure F, Jacqmin D. Natural history of residual renal stone fragments after ESWL. Eur Urol. 2000 Jan;37(1):18-22. doi: 10.1159/000020093. PMID 10671779
- [Background] Raza A, Turna B, Smith G, Moussa S, Tolley DA. Pediatric urolithiasis: 15 years of local experience with minimally invasive endourological management of pediatric calculi. J Urol. 2005 Aug;174(2):682-5. doi: 10.1097/01.ju.0000164749.32276.40. PMID 16006948
- [Background] Badawy AA, Saleem MD, Abolyosr A, Aldahshoury M, Elbadry MS, Abdalla MA, Abuzeid AM. Extracorporeal shock wave lithotripsy as first line treatment for urinary tract stones in children: outcome of 500 cases. Int Urol Nephrol. 2012 Jun;44(3):661-6. doi: 10.1007/s11255-012-0133-0. Epub 2012 Feb 16. PMID 22350835
- [Background] Rodrigues Netto N Jr, Longo JA, Ikonomidis JA, Rodrigues Netto M. Extracorporeal shock wave lithotripsy in children. J Urol. 2002 May;167(5):2164-6. PMID 11956471
- [Background] Ather MH, Noor MA. Does size and site matter for renal stones up to 30-mm in size in children treated by extracorporeal lithotripsy? Urology. 2003 Jan;61(1):212-5; discussion 215. doi: 10.1016/s0090-4295(02)02128-3. PMID 12559298
- [Background] Al-Busaidy SS, Prem AR, Medhat M. Pediatric staghorn calculi: the role of extracorporeal shock wave lithotripsy monotherapy with special reference to ureteral stenting. J Urol. 2003 Feb;169(2):629-33. doi: 10.1097/01.ju.0000047231.36474.57. PMID 12544330
- [Background] Ozgur Tan M, Karaoglan U, Sozen S, Bozkirli I. Extracorporeal shock-wave lithotripsy for treatment of ureteral calculi in paediatric patients. Pediatr Surg Int. 2003 Aug;19(6):471-4. doi: 10.1007/s00383-003-0961-1. Epub 2003 May 8. PMID 12736749
- [Background] Onal B, Demirkesen O, Tansu N, Kalkan M, Altintas R, Yalcin V. The impact of caliceal pelvic anatomy on stone clearance after shock wave lithotripsy for pediatric lower pole stones. J Urol. 2004 Sep;172(3):1082-6. doi: 10.1097/01.ju.0000135670.83076.5c. PMID 15311043
- [Background] Ozgur Tan M, Karaoglan U, Sen I, Deniz N, Bozkirli I. The impact of radiological anatomy in clearance of lower calyceal stones after shock wave lithotripsy in paediatric patients. Eur Urol. 2003 Feb;43(2):188-93. doi: 10.1016/s0302-2838(02)00492-x. PMID 12565778
- [Background] Demirkesen O, Onal B, Tansu N, Altintas R, Yalcin V, Oner A. Efficacy of extracorporeal shock wave lithotripsy for isolated lower caliceal stones in children compared with stones in other renal locations. Urology. 2006 Jan;67(1):170-4; discussion 174-5. doi: 10.1016/j.urology.2005.07.061. PMID 16413356
- [Background] Bellin MF, Renard-Penna R, Conort P, Bissery A, Meric JB, Daudon M, Mallet A, Richard F, Grenier P. Helical CT evaluation of the chemical composition of urinary tract calculi with a discriminant analysis of CT-attenuation values and density. Eur Radiol. 2004 Nov;14(11):2134-40. doi: 10.1007/s00330-004-2365-6. Epub 2004 Jun 25. PMID 15221262
- [Background] Kattan S, Husain I, el-Faqih SR, Atassi R. Incidence of bacteremia and bacteriuria in patients with non-infection-related urinary stones undergoing extracorporeal shock wave lithotripsy. J Endourol. 1993 Dec;7(6):449-51. doi: 10.1089/end.1993.7.449. PMID 8124334
- [Background] Pearle MS, Roehrborn CG. Antimicrobial prophylaxis prior to shock wave lithotripsy in patients with sterile urine before treatment: a meta-analysis and cost-effectiveness analysis. Urology. 1997 May;49(5):679-86. doi: 10.1016/S0090-4295(96)00626-7. PMID 9145970
- [Background] Leusmann DB, Tschuschke C, Stenzinger W. Extracorporeal shock wave lithotripsy of renal calculi in a patient with haemophilia A complicated by a high titre factor VIII inhibitor. Br J Urol. 1995 Mar;75(3):415-6. doi: 10.1111/j.1464-410x.1995.tb07364.x. No abstract available. PMID 7735816
- [Background] Kufer R, Thamasett S, Volkmer B, Hautmann RE, Gschwend JE. New-generation lithotripters for treatment of patients with implantable cardioverter defibrillator: experimental approach and review of literature. J Endourol. 2001 Jun;15(5):479-84. doi: 10.1089/089277901750299258. PMID 11465325
- [Background] Recker F, Hofmann W, Bex A, Tscholl R. Quantitative determination of urinary marker proteins: a model to detect intrarenal bioeffects after extracorporeal lithotripsy. J Urol. 1992 Sep;148(3 Pt 2):1000-6. doi: 10.1016/s0022-5347(17)36800-3. PMID 1507316
- [Background] Knapp PM, Kulb TB, Lingeman JE, Newman DM, Mertz JH, Mosbaugh PG, Steele RE. Extracorporeal shock wave lithotripsy-induced perirenal hematomas. J Urol. 1988 Apr;139(4):700-3. doi: 10.1016/s0022-5347(17)42604-8. PMID 3352025
- [Background] Newman LH, Saltzman B. Identifying risk factors in development of clinically significant post-shock-wave lithotripsy subcapsular hematomas. Urology. 1991 Jul;38(1):35-8. doi: 10.1016/0090-4295(91)80009-v. PMID 1866855
- [Background] Orozco Farinas R, Iglesias Prieto JI, Massarrah Halabi J, Mancebo Gomez JM, Perez-Castro Ellendt E. [Renal hematoma after extracorporeal shockwave lithotripsy in a series of 324 consecutive sessions with the DOLI-S lithotripter: incidents, characteristrics, multifactorial analysis and review]. Arch Esp Urol. 2008 Oct;61(8):889-914. doi: 10.4321/s0004-06142008000800006. Spanish. PMID 19040158
- [Background] Recker F, Rubben H, Bex A, Constantinides C. Morphological changes following ESWL in the rat kidney. Urol Res. 1989;17(4):229-33. doi: 10.1007/BF00262598. PMID 2773190
- [Background] Neuerburg J, Daus HJ, Recker F, Bohndorf K, Bex A, Guenther R, Hofstaedter F. Effects of lithotripsy on rat kidney: evaluation with MR imaging, histology, and electron microscopy. J Comput Assist Tomogr. 1989 Jan-Feb;13(1):82-9. doi: 10.1097/00004728-198901000-00018. PMID 2910952
- [Background] Delius M, Enders G, Xuan ZR, Liebich HG, Brendel W. Biological effects of shock waves: kidney damage by shock waves in dogs--dose dependence. Ultrasound Med Biol. 1988;14(2):117-22. doi: 10.1016/0301-5629(88)90178-0. PMID 3347964
- [Background] Burger W, Chemnitius JM, Kneissl GD, Rucker G. Low-dose aspirin for secondary cardiovascular prevention - cardiovascular risks after its perioperative withdrawal versus bleeding risks with its continuation - review and meta-analysis. J Intern Med. 2005 May;257(5):399-414. doi: 10.1111/j.1365-2796.2005.01477.x. PMID 15836656
- [Background] Ueda S, Matsuoka K, Yamashita T, Kunimi H, Noda S, Eto K. Perirenal hematomas caused by SWL with EDAP LT-01 lithotripter. J Endourol. 1993 Feb;7(1):11-5. doi: 10.1089/end.1993.7.11. PMID 8481715
- [Background] Oscarsson A, Gupta A, Fredrikson M, Jarhult J, Nystrom M, Pettersson E, Darvish B, Krook H, Swahn E, Eintrei C. To continue or discontinue aspirin in the perioperative period: a randomized, controlled clinical trial. Br J Anaesth. 2010 Mar;104(3):305-12. doi: 10.1093/bja/aeq003. PMID 20150346
- [Background] Ferrari E, Benhamou M, Cerboni P, Marcel B. Coronary syndromes following aspirin withdrawal: a special risk for late stent thrombosis. J Am Coll Cardiol. 2005 Feb 1;45(3):456-9. doi: 10.1016/j.jacc.2004.11.041. PMID 15680728
- [Background] Collet JP, Montalescot G, Blanchet B, Tanguy ML, Golmard JL, Choussat R, Beygui F, Payot L, Vignolles N, Metzger JP, Thomas D. Impact of prior use or recent withdrawal of oral antiplatelet agents on acute coronary syndromes. Circulation. 2004 Oct 19;110(16):2361-7. doi: 10.1161/01.CIR.0000145171.89690.B4. Epub 2004 Oct 11. PMID 15477397
- [Background] Telegrafo M, Carluccio DA, Rella L, Ianora AA, Angelelli G, Moschetta M. Diagnostic and prognostic role of computed tomography in extracorporeal shock wave lithotripsy complications. Urol Ann. 2016 Apr-Jun;8(2):168-72. doi: 10.4103/0974-7796.163792. PMID 27141186